CLINICAL TRIAL: NCT02814604
Title: FoodFLIP: Testing the Effectiveness of a Food Information App to Promote the Selection of Healthier Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Dietitians of Canada (Unknown)
Responsible Party: Principal Investigator, Mary L'Abbe, Earle W. McHenry Professor and Chair, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 499174
Record Dates: First submitted 2016-05-24; First posted 2016-06-28 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Consumer Behavior; Diet, Food, and Nutrition
Keywords: Front-of-Pack Labelling; Star rating system; Traffic light rating system; Consumer Behavior; Health Literacy; Mobile Apps; Nutrition Labeling; Healthy food choices; High-in Warning Labels
MeSH Terms: conditions — Consumer Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Traffic Light (Experimental): Participants in this group will download an app which features the nutrition information of the selected product in a multiple coloured traffic light format (i.e. the traffic light system shows a coloured round indicator for each of saturated fat, sugar, and sodium; shaded red (high), amber (medium) or green (low), according to thresholds set for each nutrient). In addition, a list of healthier similar products will appear on screen to facilitate comparisons.
  Intervention: Device:Smartphone, Behavioural: Nutrition Rating Systems
  Interventions: Other: Nutrition Rating Systems
- Health Star Rating System (Experimental): Participants in this group will download an app which features the nutrition information of the selected product in a form of 0-5 stars to provide an overall "healthy" rating. The Health Star Rating provides a rating for all products and products not meeting the criteria still carry the symbol (with no colored stars). In addition, a list of healthier similar products will appear on screen to facilitate comparisons.
  Intervention: Device:Smartphone, Behavioural: Nutrition Rating Systems
  Interventions: Other: Nutrition Rating Systems
- Control (No Intervention): Participants in this group will only see the Nutrition Facts Table (as it appears on the product's package) when the product is scanned in the app.
- High-in Warning Label (Experimental): Participants in this group will download an app which features the nutrition information of the selected product in a 'high-in' warning label format (i.e. stop signs for each of saturated fat, sugar, and sodium; according to thresholds set for each nutrient). In addition, a list of healthier similar products will appear on screen to facilitate comparisons.
  Intervention: Device:Smartphone, Behavioural: Nutrition Rating Systems
  Interventions: Other: Nutrition Rating Systems

INTERVENTIONS:
Other: Nutrition Rating Systems — Behavioural: Nutrition Rating Systems (shown on a mobile app) provide consumers with an interpretation of the healthfulness of a food or beverage product.
  Other Names: Device: Smartphone
  Arms: Health Star Rating System; High-in Warning Label; Traffic Light

SUMMARY:
There is a lot of confusion when it comes to understanding nutrition information on food packages, thus making it difficult for consumers to choose healthy products. In today's busy and fast-paced shopping environment, mobile digital technology (for example, Smartphone applications) can help consumers make 'healthier' food choices when they are shopping. This study aims to test the effectiveness of a traffic light front-of-pack system, the Health Star Rating System (HSR or Star System), and the proposed sodium, saturated fat and sugar warning labels proposed by Health Canada. The study will also experimentally test the use of a Smartphone application (app), FoodFlip, to help educate consumers on these systems on food packages to explore the impact of a learning effect on the efficacy of the labelling systems.

DETAILED DESCRIPTION:
The rising rate of obesity and diet-related chronic diseases illustrate that Canadians' eating habits need to change. Equipping Canadians with information and tools to enable healthy food choices that decrease risk for disease is imperative. While the Nutrition Facts table (NFt) is the most standardized and complete form of nutrition labelling, studies have shown that consumers are confused about serving size, nutrient quantities, and the interpretation of the % Daily Value. Thus, expert groups have proposed the introduction of interpretive front-of-pack (FOP) nutrition rating systems (e.g. traffic light labelling or star ratings) that also help consumers understand the significance of the levels of nutrients in relation to the "healthiness" of a food. One of the main barriers to the introduction of such a system is the absence of high quality studies that objectively measure the impact of nutrition information on actual food purchases. This is a consequence of both the practical challenges associated with designing and conducting such studies in 'real-world' settings, and the lack of food industry support to quantitatively examine or publish the potential for enhanced nutrition labels to modify consumer food choices. With the growing burden of diet-related disease, there is an urgent need for robust evidence to evaluate the potential for additional interpretive nutrition labelling systems to modify and improve food purchasing patterns. Given the relative ubiquity of mobile digital technologies, our Canadian Smartphone application (FoodFLIP) provides us with an unprecedented opportunity to examine and improve consumers' diets.

This study will investigate whether a traffic light, a health star rating or a high-in warning label FOP system can help consumers identify and purchase healthier foods.

Objective 1: To evaluate the effects of three FOP systems in helping consumers characterize healthfulness and nutritional content of food items.

Objective 2: To determine which of the three FOP systems support healthier food choices and are preferred by Canadian consumers.

ELIGIBILITY:
Inclusion Criteria:

* Shop at a supermarket owned by one of the largest four national retailers at least twice a month. This includes Loblaws, Sobeys, Metro or Safeway
* Own a smartphone (iPhone version 3 or later or android)
* Are 18 years or over and provide informed consent to participate
* Reside in Canada, excluding Northern Territories

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2008 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
The accurate characterization of healthfulness and nutritional content of foods as indicated by each intervention group will be compared. | 6 weeks
  In the first series of experimental tasks, participants will be exposed to an image of a food package with the assigned FOP nutrition information and NFt. Participants will be asked to rate the products on how likely they would be to purchase the product, overall healthiness, and the relative amount of specific nutrients in the product (e.g., if the product contains a little or a lot of sodium) using a Likert scale. In the second series of tasks, participants will be shown 5 similar products side by side (5 breakfast cereals, 5 yogurts and 5 pasta dinners). Participants will be asked to rank the products from MOST HEALTHY to LEAST HEALTHY, and which product they would select if they were trying to consume a low sodium, low energy or high fibre diet.

SECONDARY OUTCOMES:
A qualitative assessment of the functionality and usability of the smartphone app (FoodFLIP) will be assessed through questionnaires on a 5-point Likert Scale (the percentage of users finding the app easy to use/easy to understand etc). | 6 weeks
  The functionality and usability of the smartphone app is assessed through questionnaires (e.g easy to use, easy to understand etc). Responses on these questionnaires are scaled using a five-point Likert-scale and scores for each question are recorded separately to assess the usability of the smartphone app (e.g 1 least liked to 5 most liked).
The health claims with or without additional labelling elements influence perceptions of healthiness and purchasing intentions will be compared between each FOP system. | 6 weeks
  Participants will be randomized to see products with symbolic and textual health and/or nutrition claims. Participants will first be shown an image with or without claims for 10 seconds (this is slightly longer than the average time an individual spends viewing a product in a food store when making a purchasing decision). The image will then be removed from the screen, and participants will be asked to recall the presence and content of the claim. The image will then be returned to the screen and participants will be asked to rate how healthy the product is and to rate how likely they would be to purchase the product.

CONTACTS AND LOCATIONS:
Overall Officials: Mary R L'Abbe, Ph.D., Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Key TJ, Schatzkin A, Willett WC, Allen NE, Spencer EA, Travis RC. Diet, nutrition and the prevention of cancer. Public Health Nutr. 2004 Feb;7(1A):187-200. doi: 10.1079/phn2003588. PMID 14972060
- [Background] Emrich TE, Qi Y, Mendoza JE, Lou W, Cohen JE, L'abbe MR. Consumer perceptions of the Nutrition Facts table and front-of-pack nutrition rating systems. Appl Physiol Nutr Metab. 2014 Apr;39(4):417-24. doi: 10.1139/apnm-2013-0304. Epub 2013 Oct 24. PMID 24669982
- [Background] The Standing Committee on Health. Healthy Weights for Healthy Kids. 2007
- [Background] McGuire S. Institute of Medicine. 2012. Front-of-Package Nutrition Rating Systems and Symbols: Promoting Healthier Choices. Washington, DC: The National Academies Press. Adv Nutr. 2012 May 1;3(3):332-3. doi: 10.3945/an.112.001933. No abstract available. PMID 22585907